CLINICAL TRIAL: NCT05271357
Title: Theta Burst Stimulation for Refractory Depression in Autism Spectrum Conditions
Brief Title: Transcranial Magnetic Stimulation for Depression in Autism Spectrum Conditions
Acronym: RESTORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Ernest Pedapati, MD, Associate Professor, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0594
Record Dates: First submitted 2021-10-28; First posted 2022-03-09 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Autism Spectrum Disorder; Major Depressive Disorder
Keywords: Transcranial magnetic stimulation; TMS; MDD; ASD; TBS; theta burst stimulation; autism; depression
MeSH Terms: conditions — Autism Spectrum Disorder; Depressive Disorder, Major; Autistic Disorder; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bilateral (Experimental): Theta burst stimulation (TBS)
  Interventions: Procedure: Bilateral TMS
- Unilateral (Active Comparator): Theta burst stimulation (TBS)
  Interventions: Procedure: Unilateral TMS

INTERVENTIONS:
Procedure: Bilateral TMS — Stimulation begins with continuous TBS to the right dorsolateral prefrontal cortex (DLPFC) (120 seconds of uninterrupted bursts; 600 pulses per session) followed by intermittent TBS to the left DLPFC (2 seconds on and 8 seconds off; 600 pulses per session); total duration of 3 min 9 seconds per hemisphere.
  Arms: Bilateral
Procedure: Unilateral TMS — Stimulation involves only intermittent TBS to the left DLPFC (2 seconds on and 8 seconds off; 600 pulses per session); total duration of 3 min 9 seconds.
  Arms: Unilateral

SUMMARY:
In this research study the investigators aim to learn more about the therapeutic effects of a newer form of non-invasive transcranial magnetic stimulation (TMS), called theta burst simulation (TBS), on refractory depression in Autism Spectrum Conditions.

DETAILED DESCRIPTION:
The overarching goal of this study is to examine treatment effects and elucidate the physiological biomarkers of a newer form of non-invasive brain stimulation therapy on refractory depression in a sample of participants with ASC (autism spectrum condition).

Aim 1: To compare the efficacy of 30-sessions of bilateral (BL) versus unilateral (UL) Theta Burst Stimulation to the dorsolateral prefrontal cortex (DLPFC) on depression severity in youth/young adults with ASC and co-occurring refractory major depressive disorder (MDD).

Aim 2: To identify physiological markers of target engagement of successful response to either UL or BL on depression severity in youth with ASC and co-occurring refractory MDD. These physiological markers include high-resolution electroencephalography (EEG) markers, social eye-tracking, and handgrip strength (collected via NIH toolbox's motor toolbox domain).

Aim 3: To identify feasibility of BL and UL in participants with ASC including systematic measures of safety and tolerability. This includes clinical measures such as rate of hospitalization and medication use.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed on the autism spectrum
* Have been diagnosed with depression and have failed one or more evidence-based antidepressant treatments (e.g. a Selective Serotonin Reuptake Inhibitor, talk therapy like Cognitive Behavioral Therapy)
* Do not have an intellectual disability

Exclusion Criteria:

* Substance use disorder
* Presence of metallic foreign bodies or implanted medical devices
* History of epilepsy
* Prior rTMS treatment
* For female subjects of child bearing potential, current pregnancy

Ages: 12 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Change-from-baseline at 4 weeks in mean Hamilton Depression Rating Scale (HDRS-17) score. | 4 weeks post-treatment
  The HDRS-17 is a valid and reliable measure that assesses severity of, and change in, depressive symptoms. HDRS-17 scores range from 0-52, with scores of 0-7 indicating absence or remission of depression, 7-17 indicating mild depression, 18-24 indicating moderate depression, and scores at or over 25 indicating severe depression.
Change-from-baseline at 4 weeks in mean and Beck Depression Inventory (BDI-II) scores. | 4 weeks post-treatment
  The BDI-II is a valid and reliable measure for assessing the severity of depressive symptoms. BDI-II scores range from 0-63, with scores of 0-10 indicating absence or remission of depression, 11-16 indicating mild mood disturbance, 17-20 indicating borderline clinical depression, 21-30 indicating moderate depression, 31-40 severe depression, and scores over 40 indicating extreme depression.

SECONDARY OUTCOMES:
Change-from-baseline at 4 weeks in physiological markers via the use of high-resolution electroencephalography (EEG). | 4 weeks post-treatment
  EEG offers a real-time image of cortical excitability and connectivity. We will use power spectral analysis to assess changes in event-related gamma and alpha activity.
Change-from-baseline at 4 weeks in handgrip strength or relative handgrip strength. | 4 weeks post-treatment
  Handgrip strength is particularly novel and has been shown to be negatively associated with depressive symptoms, making muscle strength a possible clinical marker of poor mental health. The grip strength test from NIH Toolbox's motor domain will be used to collect a digital reading of force in pounds from each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Pedapati, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: upon completion of data collection

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT05271357/Prot_SAP_002.pdf